CLINICAL TRIAL: NCT04906291
Title: The Caries Preventive Effect of 2-years Use of Hydroxyapatite Containing Toothpastes in Children. A Triple-blind Randomized Placebo-controlled Clinical Trial.
Brief Title: The Preventive Effect of 2-years Use of Hydroxyapatite Containing Toothpastes in Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Guglielmo Campus, Associate Professor in Preventive Dentistry, Università degli Studi di Sassari
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: USassari02.2017
Record Dates: First submitted 2021-05-24; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Caries
Keywords: Toothpaste, hydroxyapatite, Fluoride, Dental Caries, RCT, Children
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- H.A.F. toothpaste (1000 ppm F-) (Experimental): The children were instructed to brush their teeth for at least two minutes after each main meal (three times/day).
  Interventions: Other: Toothpaste use
- Fluoridated toothpaste (1000 ppm F-) (Active Comparator): The subjects were instructed to brush their teeth for at least two minutes after each main meal (three times/day).
  Interventions: Other: Toothpaste use
- H.A.F. toothpaste (1450 ppm F-) (Experimental): The subjects were instructed to brush their teeth for at least two minutes after each main meal (three times/day).
  Interventions: Other: Toothpaste use
- Fluoridated toothpaste (1450 ppm F-) (Active Comparator): The subjects were instructed to brush their teeth for at least two minutes after each main meal (three times/day).
  Interventions: Other: Toothpaste use

INTERVENTIONS:
Other: Toothpaste use — Brushing three times a day

SUMMARY:
The aim of this RCT was to verify the caries preventive efficacy of toothpastes containing biomimetic hydroxyapatite (H.A.) complex in children compared to traditional fluoridated toothpastes. In total 610 children of two age groups (4-5 years and 6-7 years at baseline) were enrolled. Four toothpastes, two containing fluoride-substituted hydroxyapatite (H.A.F.) (1000 and 1450 ppm F-) and magnesium-, strontium-, carbonate-substituted hydroxyapatite, in a chitosan matrix and two traditional fluoridated toothpastes (1000 and 1450 ppm F-) without other active components were administered randomly to two groups with younger children (Gyoung) and to two groups with older children those containing1450 ppm F (GOLD) during 24 months. A standardized questionnaire was administered to parents/caregivers to gain information regarding caries risk factors. Caries evaluation was performed at school using ICDAS, scoring lesions as initial (up to score 2), moderate (scores 3-4) and severe (scores 5-6).

ELIGIBILITY:
Inclusion Criteria:

* Written declaration of informed consent signed by parents/guardians;
* Age between 4-5 years and 6-7 years; Good general health, as assessed by the examiners;
* Agreement of not to use any oral hygiene products except for the toothpastes provided for the duration of the study.

Exclusion Criteria:

* Ongoing oral or dental treatment except for emergency treatment;
* Known allergic reaction to an oral hygiene product and/or medication and/or dental material previously used in the mouth or pharynx;
* Allergy to one of the components of the test products or the standard toothpaste;
* Participation in another clinical trial either currently or within the last 30 days;
* Antibiotic therapy within the past 3 months.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 610 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Caries Progression rate | 2 year
  . Caries incidence rate was calculated on each tooth (primary and permanent) as the unit of analysis

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sassari, Dept of Surgery, Microsurtgery and Medicine Sciences, Sassari, SS, Italy

IPD SHARING:
Plan to Share IPD: No